CLINICAL TRIAL: NCT05130138
Title: Interest of PHARMaceutical Conciliation to Understand Drug Interactions, Phytotherapy, and Targeted Therapies in Chronic Myeloid Leukemia: PHARM-LMC Study
Brief Title: Interest of PHARMaceutical Conciliation to Understand Drug Interactions, Phytotherapy, and Targeted Therapies in Chronic Myeloid Leukemia
Acronym: PHARM-LMC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-0401; 2021-A00942-39 (Other: Agence Nationale de Sécurité du Médicament et des produits de santé)
Record Dates: First submitted 2021-10-13; First posted 2021-11-22 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Chronic Myeloid Leukemia
Keywords: hematology; Chronic Myeloid Leukemia; Tyrosine Kinase Inhibitor; pharmaceutical conciliation; pharmaceutical intervention; drug interactions; phytotherapy; targeted therapies
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pharmaceutical conciliation (Experimental): Patients with Chronic Myeloid Leukemia taking TKI with a molecular response < 4,5 Log will participate to pharmaceutical conciliation.
  Interventions: Other: Pharmaceutical intervention

INTERVENTIONS:
Other: Pharmaceutical intervention — Patients with pharmacokinetic and/or pharmacodynamics interactions will be proposed to participate to educational sessions to discuss about treatments taken and modifications possibilities.

SUMMARY:
The aim of this trial is therefore to identify concomitant treatments with taking Tyrosine Kinase Inhibitor (=TKI) in the indication of Chronic Myeloid Leukemia (CML), whatever the stage of the disease, via pharmaceutical conciliation. These concomitant treatments as well as their dosages will be correlated with the TKI dosage since patients must have a sufficient residual concentration to be considered effective and to confirm adherence to treatment, the leading cause of treatment failure.

In the event of unsatisfactory results, pharmaceutical interventions may take place: changes in treatments (TKI and not TKI) and / or dosages. In case of modification, a new dosage of TKI should be carried out.

DETAILED DESCRIPTION:
Chronic myeloid leukemia (CML) is a clonal myeloproliferative syndrome with an estimated incidence of 0.8-1 cases per 100,000 person-years in 2018 in France. CML is characterized by the transformation of a pluripotent stem cell resulting in an increase in myeloid and erythroid lineages and megakaryocytes in peripheral blood as well as myeloid hyperplasia in the bone marrow.

In the absence of treatment, the disease, which begins in a chronic phase over a few years, progresses to an acceleration phase, before reaching an acute phase, known as a blast crisis, with a poor prognosis. This abnormal proliferation of white blood cells results from the reciprocal translocation (exchange) between chromosomes 9 and 22. This exchange brings two normally distinct genes into contact: the (breakpoint cluster region) BCR gene and the abl gene (Tyrosine-protein kinase), which will form an abnormal gene called "fusion Bcr-abl". This gene encodes a fusion protein with deregulated tyrosine kinase activity that activates various mechanisms involved in cell multiplication.

Since the 1990s, the arrival of the first tyrosine kinase inhibitor (TKI), imatinib, has radically changed patient management. Indeed, according to Public Health France, this treatment has allowed the majority of patients to remain in the chronic phase for a long time. Patient survival has therefore increased dramatically as the life expectancy of patients with CML taking their treatment regularly approaches that of the general population.

However, even though several generations of TKI have been developed, certain toxicities may lead to discontinuation of treatment, or to a modification of the dose. Indeed, a meta-analysis published in June 2020 shows that second and third generation of TKI improve the major molecular response by 3 months, but are associated with a recrudescence of thrombocytopenia, cardiovascular, pancreatic and hepatic events. First generation imatinib therefore remains the best option for patients with co-morbidities despite the frequent presence of headaches, digestive disorders, and cramps.

It has therefore always been customary to change the TKI or modify the prescribed doses, while the side effects or ineffectiveness of these inhibitors could be explained by drug interactions, or be related to the use of herbal medicine. Indeed, TKIs are metabolized by the cytochrome P450 system. The activity of this cytochrome is not only different from one person to another, but can also be affected by other treatments. For example, some treatments will inhibit the activity of this cytochrome P450, increasing the exposure of TKIs in plasma. The pharmacokinetics of the drug will therefore depend on these concomitant treatments and their influence, among others, on cytochrome P450.

In addition, the median age at diagnosis is respectively 61 years for men and 62 years for women. These patients are therefore often carriers of other chronic diseases and are have multiple treatments.

ELIGIBILITY:
Inclusion Criteria:

* Major patient;
* Patient affiliated to a social security scheme;
* Patient suffering from Chronic Myeloid Leukemia, taking a Tyrosine Kinase Inhibitor (Imatinib, Nilotinib, Dasatinib, or Bosutinib);
* Molecular response < 4,5 Log;

Exclusion Criteria:

* Legal incapacity or limited capacity ; Medical or psychological incapacity or limited capacity;
* Not able to read and/or to write French;
* Patient taking Ponatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients for whom pharmaceutical interventions have been done | 12 months
  Number of patients for whom pharmaceutical interventions have been done secondly to pharmaceutical conciliation will be reported.

SECONDARY OUTCOMES:
Molecular response | 12 months
  Molecular response will be reported via BCR-ABL transcript rate measured by quantitative polymerase chain reaction (qPCR) or digital polymerase chain reaction (PCR).
Concomitant treatments | 12 months
  Concomitant treatments will be reported during 12 months.
Tyrosine kinase inhibitor observance | 12 months
  Observance to Tyrosine kinase inhibitor will be measured with Girerd Questionnaire.
Side effects | 12 months
  Number and description of sides effects will be reported.
Patients' satisfaction | 12 months
  Patients' satisfaction will be measured with a visual scale from 0 to 10.
Patients' quality of life | 12 months
  Patients' quality of life will be measured with the Quality of Life questionnaires (QLQ-C30) questionnaire. The maximum score is 126, the minimum score is 30. More the score is, worst the health state is.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier SIMOENS, MD, PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No